CLINICAL TRIAL: NCT00506636
Title: Study of Tissue Engineering for Hair Follicle Regeneration
Brief Title: Tissue Engineering for Hair Follicle Regeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Other Study IDs: 9561705025
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2006-05

CONDITIONS: Tissue Engineering; Hair Follicle Regeneration
MeSH Terms: interventions — Tissue Engineering

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Tissue engineering for hair follicle regeneration

SUMMARY:
This study is to try to maintain cultured dermal papilla cells in spherical structure in vitro before transplanting into dermis in vivo. Also, this study is aimed in clarifying actual mechanism of inducing hair follicle by dermal papilla cells.

DETAILED DESCRIPTION:
Hair transplantation is an well-documented way of treating hair loss. Hair transplantation is based on redistribution of hair follicles without any new follicle formation. It has been long that a lot of researchers have focused on developing skills in regenerating hair follicles. However, cultured dermal papilla cells lose the ability of inducing hair follicle formation after several generations in vitro culture. Our study is aiming in culturing dermal papilla cells in vitro and maintain their spherical structure before transplanting into dermis in vivo. Meantime, this study may help clarify the actual mechanism of inducing hair follicle by dermal papilla cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving cosmetic surgeries such as removal of moles

Exclusion Criteria:

* No special exclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-05; Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Jan Lin, MD PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan